CLINICAL TRIAL: NCT05928806
Title: Phase 2 Advanced Renal Cell Cancer Combination ImmunoThErapy Clinical Trial
Brief Title: Advanced Renal Cell Cancer Combination ImmunoThErapy Clinical Trial
Acronym: ARCITECT
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim Analysis
Sponsor: Michael B. Atkins, MD (Other)
Collaborators: Agenus Inc. (Industry); Georgetown University (Other)
Responsible Party: Sponsor-Investigator, Michael B. Atkins, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU22-587
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Renal Cell Carcinoma
MeSH Terms: interventions — balstilimab; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (botensilimab and balstilimab) (Experimental): Arm A subjects will receive 2 cycles of induction treatment with each cycle lasting 6 weeks. Cycle 1 will consist of botensilimab 75mg IV in combination with balstilimab 450mg IV on Day 1 and Day 22. Cycle 2 will consist of balstilimab 450mg IV ONLY on Day 1 and Day 22. Botensilimab will NOT be given in Cycle 2. Subjects will receive 7 cycles of maintenance treatment with each cycle lasting 12 weeks. Cycles 3 and 4 will consist of botensilimab 75mg IV on Day 1 in combination with balstilimab 450mg IV on Day 1, 22, 43 and 64. Cycles 5-9 will consist of balstilimab alone 450 mg IV on Day 1, 22, 43 and 64.
  Interventions: Drug: Botensilimab; Drug: Balstilimab
- Arm B (ipilimumab and nivolumab) (Active Comparator): Arm B subjects will receive 2 cycles of induction treatment with each cycle lasting 6 weeks. Cycle 1 and 2 will consist of ipilimumab 1 mg/kg IV and nivolumab 3 mg/kg on Day 1 and 22. Subjects will receive 7 cycles of maintenance treatment with each cycle lasting 12 weeks. Nivolumab 480mg IV will be given on Day 1, 29 and 57 of each cycle (every 4 weeks).
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Botensilimab — Botensilimab 75mg IV
  Other Names: AGEN1181
  Arms: Arm A (botensilimab and balstilimab)
Drug: Balstilimab — Balstilimab 450mg IV
  Other Names: AGEN2034
  Arms: Arm A (botensilimab and balstilimab)
Drug: Ipilimumab — Ipilimumab 1mg/kg IV
  Other Names: Yervoy
  Arms: Arm B (ipilimumab and nivolumab)
Drug: Nivolumab — Nivolumab at induction: 3mg/kg IV Nivolumab at maintenance: 480mg IV
  Other Names: Opdivo
  Arms: Arm B (ipilimumab and nivolumab)

SUMMARY:
This study is a randomized, open label, multicenter Phase II trial to evaluate the efficacy and safety of botensilimab (a novel Fc enhanced Tree depleting anti-CTLA4) and balstilimab (a novel anti-PD1) relative to ipilimumab and nivolumab in treatment naïve patients with metastatic ccRCC. The study will plan to enroll 120 eligible patients randomized in a 2:1 fashion to Arm A and Arm B. Patients in all IMDC Risk Groups are included. This study utilizes a Simon's two stage design which is described in the protocol. Patients randomized to Arm A will receive botensilimab in combination with balstilimab. Patients randomized to Arm B will receive ipilimumab in combination with nivolumab. Study treatment on both arms will continue until toxicity, disease progression or a maximum of 96 total weeks (12 weeks induction, 84 weeks maintenance).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have ECOG PS of ≤ 2 within 28 days of C1D1.
2. Age ≥ 18 years old at the time of informed consent.
3. Patient must have histological confirmation of renal carcinoma with clear cell component including advanced RCC (not amenable to curative surgery or radiation therapy) or metastatic RCC.
4. Patient must have measurable disease by CT or MRI per RECIST 1.1 criteria. Radiated lesions cannot be used as measurable lesions unless there is clear evidence of progression.
5. Patient must have defined IMDC risk categorization of either favorable, intermediate or poor based on clinical variables of increased risk (below).

   * No risk factors (0) = favorable risk
   * 1-2 risk factors = intermediate risk
   * ≥ 3 risk factors = poor risk

   NOTE: Patients with all IMDC risk factors are eligible, but will be stratified according to IMDC risk, and initial analysis will be based on the IMDC intermediate and poor risk patients. IMDC Risks:
   * KPS less than 80%
   * Less than 1 year from diagnosis including original localized disease to randomization(if applicable)
   * Hemoglobin less than the lower limit of normal
   * Corrected calcium concentration greater than 10 mg/dL
   * ANC greater than the ULN
   * Platelet count greater than the ULN
6. Patient must have either a formalin-fixed, paraffin-embedded (FFPE) tissue block or at least 10 (preferably 20) unstained tumor tissue sections, obtained from a metastatic lesion, preferably within 3 months or no more than 12 months with an associated pathology report. This tissue must be identified prior to registration. Confirmation of sufficient archival tissue must be obtained after informed consent and the tissue must be shipped to the appropriate lab by end of Cycle 2. Biopsies should be excisional, incisional, or core needle. Fine needle aspiration is unacceptable for submission. Biopsies of bone lesions that do not have a soft tissue component are also unacceptable for submission. This sample is required to be eligible for the trial. If a patient is having a standard of care biopsy, part of that sample may be utilized for eligibility.
7. Demonstrate adequate organ function as defined below; all screening labs to be obtained within 28 days prior to registration.

   * Hematological
   * White blood cell (WBC) ≥ 2,000/uL
   * Absolute Neutrophil Count (ANC) ≥ 1,000/uL; without growth factor support
   * Hemoglobin (Hgb) ≥ 8.0 g/dL; ≥ 7 days without PRBC transfusion.
   * Platelets ≥ 75,000/uL; without platelet transfusion
   * Renal
   * Calculated creatinine clearance (CrCl)1 ≥ 40 mL/min
   * Hepatic
   * Total Bilirubin ≤ 1.5 × upper limit of normal (ULN) *EXCEPT participants with Gilbert Syndrome who must have a Total Bilirubin level of < 3.0 x ULN
   * Aspartate aminotransferase (AST) ≤ 3.0 × ULN
   * Alanine aminotransferase (ALT) ≤ 3.0 × ULN
8. HIV positive patients may be eligible if either:

   * Patients with CD4 > 200 cells/mm3 OR
   * Patients with HIV viral load undetectable.
9. Active HBV or active HCV patients may be eligible if:

   * Patients with HBV infection are eligible if hepatitis B surface antigen and HBV DNA are negative.
   * Patients with HCV infection are eligible if HCV RNA is negative.
10. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 1 week prior to Cycle 1 Day 1.
11. WOCBP must agree to follow instructions for method(s) of contraception.
12. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception.

Exclusion Criteria:

1. Prior adjuvant or systemic therapy for RCC.
2. Prior treatment with an anti-PD1 or anti-PDL1 agent, anti-CTLA4 antibody or a VEGFR TKI or anti-VEGF antibody including in the adjuvant setting.
3. Radiotherapy within 2 weeks prior to Cycle 1 Day 1.
4. Expected to require any other form of systemic or localized antineoplastic therapy while on trial (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
5. Currently known active and definitive CNS metastases. Patients who have treated brain metastases (with either surgical resection or stereotactic radiosurgery (SRS)) may be eligible. Patients must not have taken any steroids ≤ 2 weeks prior to randomization for the purpose of managing their brain metastases. Repeat imaging after SRS or surgical resection is not required so long as baseline MRI is within 4 weeks of registration. Patients with multiple brain metastases treated with SRS (with or without WBRT), are not excluded. Patients with definitive CNS metastases treated with only WBRT are ineligible. Patients with potential CNS metastases that are too small for treatment with either SRS or surgery (e.g. 1-2 mm) and/or are of uncertain etiology are potentially eligible, but need to be discussed with and approved by the sponsor-investigator.
6. Persistent toxicity of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grade > 1 severity that is related to prior therapy. NOTE: Sensory neuropathy or alopecia of Grade ≤ 2 are acceptable.
7. Known severe (Grade ≥ 3) hypersensitivity reactions to fully human monoclonal antibodies, antibody, or severe reaction to immuno-oncology agents, such as colitis or pneumonitis requiring treatment with steroids; or has a history of interstitial lung disease, any history of anaphylaxis, or uncontrolled asthma.
8. Known condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses <10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. NOTE: Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed.
9. Active known or suspected autoimmune disease that required systemic treatment within 2 years of the start of study drug (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (e.g., celiac disease) are permitted to enroll.
10. Uncontrolled adrenal insufficiency based on investigator discretion.
11. Active infection requiring systemic therapy within 14 days of Cycle 1 Day 1.
12. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 6 months of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ II), or serious uncontrolled cardiac arrhythmia requiring medication.
13. Legally incapacitated or has limited legal capacity.
14. Pregnant or breastfeeding.
15. Prior allogeneic tissue/solid organ transplant, except for corneal transplants.
16. Major surgery (e.g., nephrectomy) less than 28 days prior to Cycle 1 Day 1.
17. Prior malignancy active within the previous 2 years from screening except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
18. Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator, would preclude the participant from adhering to the protocol or would increase the risk associated with study participation or study treatment administration or interfere with the interpretation of safety results.
19. Receipt of a live/attenuated vaccine within 30 days of first study treatment. The use of inactivated seasonal influenza vaccines (eg, Fluzone®) will be permitted on study without restriction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-11-10 (Estimated)

PRIMARY OUTCOMES:
Determine the objective response rate (ORR) of botensilimab + balstilimab in patients with treatment naïve metastatic ccRCC relative to the ORR of patients treated with ipilimumab + nivolumab. | 5 years
  ORR is defined as the proportion of the subjects in the analysis population who have a CR or PR per RECIST 1.1.

SECONDARY OUTCOMES:
Determine Duration of response (DOR) for patients who have a CR or PR | 5 years
  DOR is defined as the time from first documented evidence of CR or PR per RECIST 1.1 until disease progression based on RECIST 1.1 or death due to any cause, whichever occurs first.
Determine the 12- & 24-month landmark progression free survival (PFS) | 5 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first.
Determine treatment free survival (TFS) | 5 years
  TFS will be assessed based on the area between two time to event KM curves. 1. time from study treatment initiation to study treatment discontinuation (last dose + dosing interval). 2. Time from study initiation to initiation of subsequent systemic anti-cancer treatment or death. Time on or off treatment with Grade 3 or greater treatment related toxicities per CTCAE v5 will be determined as the area between study initiation and toxicity start and study initiation and Grade 3 toxicity ending.
Determine the safety of botensilimab + balstilimab relative to ipilimumab + nivolumab | 5 years
  AEs and SAEs graded per NCI CTCAE v5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Atkins, MD, Principal Investigator — Georgetown University
Locations (13):
- United States (13):
  - University of California San Diego, La Jolla, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber - Partners Cancer Care, Inc, Boston, Massachusetts
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Cornell University, Ithaca, New York
  - Columbia University Irving Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn Medicine Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas